CLINICAL TRIAL: NCT03954535
Title: Preventing Drug Abuse Among Sexual-Minority Youth
Brief Title: Preventing Drug Abuse Among Sexual Minority Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Traci M. Schwinn, Research Scientist in the Faculty of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAR5072; R01DA043512 (NIH)
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Substance Abuse
Keywords: sexual minorities; prevention; web-based intervention; substance use; longitudinal; randomized controlled trial; adolescence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 9 sessions and website with entertainment features and resources
  Interventions: Behavioral: Free2b
- Control (Placebo Comparator): website with entertainment features and resources
  Interventions: Behavioral: Attention-Placebo

INTERVENTIONS:
Behavioral: Free2b — The intervention will consist of a website and 9 sessions. The intervention sessions will facilitate youths' acquisition of personal and social cognitive-behavioral skills. The intervention will focus on goal setting, decision making, enhancing self-worth, coping with stress, combating distorted thinking, communication skills, using alcohol and other drugs and a review session. Each session will require approximately 20 minutes and must be finished in a single sitting. Sessions will be delivered on a weekly basis. The website will include entertainment features and resources.
  Arms: Intervention
Behavioral: Attention-Placebo — Access to the website with entertainment features and resources - but no session content.
  Arms: Control

SUMMARY:
The planned randomized clinical trial will longitudinally test a tailored, web-based drug abuse prevention program with a nationwide sample of 15- to 17-year-old sexual minority youth (youth who identify as gay, lesbian, bisexual, or unsure of their sexual orientation).

DETAILED DESCRIPTION:
The randomized controlled trial will include at least 890 sexual-minority youth from the United States. Study participants will be 15- to 17-year-old youth recruited from Facebook/Instagram. All youth will complete pretest measures online. Intervention-arm youth will then interact with the 9-session program; youth in the control arm will have access to an attention-placebo website. All youth will then complete posttest measures (immediately following intervention completion and estimated to be approximately 5 months after study onset) and 1-, 2-, and 3-year follow-up measures.

Across posttest and annual follow-up measurement occasions, data analyses will examine rates of 30-day drug use between study arms. The investigators will also examine intervention effects on mediator variables associated with drug use and assess the extent to which changes in mediator variables explain differences in drug use between arms.

Youth assigned to the intervention arm will have access to 9 intervention sessions delivered online. The sessions will be housed on a website with entertainment features youth seek: life hacks, features on LGBTQ leaders, fortunes, horoscopes, inspiring quotes, and health-related resources.

To ensure that youths' expectations for study participation are equivalent across arms and to account for the non-active components of the experimental intervention, the investigators designed the attention-placebo arm. Youth assigned to the attention-placebo arm will have access to the website with entertainment features: life hacks, features on LGBTQ leaders, fortunes, horoscopes, inspiring quotes, and health-related resources.

ELIGIBILITY:
Inclusion Criteria:

* teenagers between the ages of 15-17 years old
* identify as lesbian, gay, bisexual, or unsure of sexual orientation
* speak and read English
* access to a private desktop, laptop, or tablet with broadband internet access

Exclusion:

- Lives outside the United States of America

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1216 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Traci M. Schwinn, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weisblum M, Trussell E, Schwinn T, Pacheco AR, Nurkin P. Screening and Retaining Adolescents Recruited Through Social Media: Secondary Analysis from a Longitudinal Clinical Trial. JMIR Pediatr Parent. 2024 Feb 28;7:e47984. doi: 10.2196/47984. PMID 38416559

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention-Placebo Control: website with entertainment features and resources
  Attention-Placebo: Access to the website with entertainment features and resources - but no session content.
Period: Overall Study
Arm/Group | Intervention | Attention-Placebo Control
Started | 608 | 608
Completed | 574 | 602
Not Completed | 34 | 6

BASELINE CHARACTERISTICS:
Population: 8 participants did not complete baseline assessments. Baseline data was not collected from these participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 602 | 606 | 1208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 602 | 606 | 1208
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.15 (0.57) | 16.16 (0.56) | 16.16 (0.56)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Female | 339 | 331 | 670
  Gender Identity: Male | 107 | 113 | 220
  Gender Identity: Transgender | 28 | 32 | 60
  Gender Identity: Non-binary | 74 | 73 | 147
  Gender Identity: Gender fluid | 24 | 18 | 42
  Gender Identity: Not sure | 30 | 39 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 112 | 227
  Not Hispanic or Latino | 482 | 492 | 974
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 10 | 16
  Asian | 43 | 34 | 77
  Native Hawaiian or Other Pacific Islander | 5 | 5 | 10
  Black or African American | 39 | 56 | 95
  White | 341 | 373 | 714
  More than one race | 163 | 126 | 289
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 602 | 606 | 1208

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Times Youth Drank Alcohol in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: The analyzed population reflects only those participants who completed the assessment at approx. 5 months after baseline.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 605
number of times | 0.83 (2.12) | 1.03 (2.26)

2. Primary Outcome: Average Number of Times Youth Drank Alcohol in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 603
number of times | 1.22 (2.49) | 1.37 (2.64)

3. Primary Outcome: Average Number of Times Youth Drank Alcohol in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 566 | 596
number of times | 1.93 (3.91) | 2.30 (4.74)

4. Primary Outcome: Average Number of Times Youth Drank Alcohol in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 572 | 598
number of times | 2.49 (4.86) | 2.67 (5.72)

5. Primary Outcome: Average Number of Times Youth Binge Drank in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 604
number of times | 0.18 (0.88) | 0.25 (0.97)

6. Primary Outcome: Average Number of Times Youth Binge Drank in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 602
number of times | 0.35 (1.05) | 0.32 (0.97)

7. Primary Outcome: Average Number of Times Youth Binge Drank in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 595
number of times | 0.50 (1.38) | 0.59 (1.60)

8. Primary Outcome: Average Number of Times Youth Binge Drank in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 571 | 597
number of times | 0.65 (1.64) | 0.78 (2.41)

9. Primary Outcome: Average Number of Times Youth Smoked Cigarettes in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 605
number of times | 0.31 (3.23) | 0.39 (4.29)

10. Primary Outcome: Average Number of Times Youth Smoked Cigarettes in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 602
number of times | 0.50 (4.11) | 0.48 (3.74)

11. Primary Outcome: Average Number of Times Youth Smoked Cigarettes in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 596
number of times | 0.70 (5.23) | 0.79 (5.67)

12. Primary Outcome: Average Number of Times Youth Smoked Cigarettes in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year-follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 572 | 597
number of times | 0.76 (5.27) | 1.05 (6.61)

13. Primary Outcome: Average Number of Times Youth Smoked Marijuana in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 565 | 604
number of times | 2.43 (10.23) | 1.89 (7.54)

14. Primary Outcome: Average Number of Times Youth Smoked Marijuana in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 599
number of times | 4.64 (13.67) | 3.71 (12.03)

15. Primary Outcome: Average Number of Times Youth Smoked Marijuana in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 564 | 595
number of times | 7.12 (17.53) | 7.04 (17.07)

16. Primary Outcome: Average Number of Times Youth Smoked Marijuana in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 593
number of times | 8.53 (17.99) | 8.54 (17.97)

17. Primary Outcome: Average Number of Times Youth Vaped Any Substance in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 566 | 604
number of times | 3.09 (11.69) | 2.95 (11.24)

18. Primary Outcome: Average Number of Times Youth Vaped Any Substance in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 596
number of times | 6.60 (17.47) | 5.80 (16.13)

19. Primary Outcome: Average Number of Times Youth Vaped Any Substance in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 566 | 594
number of times | 9.23 (20.68) | 9.87 (21.33)

20. Primary Outcome: Average Number of Times Youth Vaped Any Substance in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 594
number of times | 11.99 (23.28) | 11.11 (22.32)

21. Primary Outcome: Average Number of Times Youth Used Hard Drugs in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 565 | 604
number of times | 0.65 (3.63) | 0.71 (4.35)

22. Primary Outcome: Average Number of Times Youth Used Hard Drugs in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 599
number of times | 0.58 (3.92) | 0.60 (3.84)

23. Primary Outcome: Average Number of Times Youth Used Hard Drugs in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 564 | 598
number of times | 0.45 (2.67) | 0.61 (4.34)

24. Primary Outcome: Average Number of Times Youth Used Hard Drugs in the Past Month
Description: Participants will be asked to report the numbers of times they have used the substance in the past month.
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 593
number of times | 0.34 (1.92) | 0.62 (3.65)

25. Secondary Outcome: Mean Scores for Goal Setting
Description: The goal setting scale is a 5-item measure assessing the degree to which youth set and work on goals. All items are averaged to yield a total score that ranges from 0 = low goal setting to 3 = higher goal setting; higher scores indicate a better outcome. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 603
score on a scale | 2.38 (0.60) | 2.34 (0.62)

26. Secondary Outcome: Mean Scores for Goal Setting
Description: as for outcome 25
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 602
score on a scale | 2.39 (0.63) | 2.36 (0.61)

27. Secondary Outcome: Mean Scores for Goal Setting
Description: as for outcome 25
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 595
score on a scale | 2.47 (0.63) | 2.39 (0.63)

28. Secondary Outcome: Mean Scores for Goal Setting
Description: as for outcome 25
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 596
score on a scale | 2.57 (0.65) | 2.49 (0.62)

29. Secondary Outcome: Mean Scores for Problem Solving
Description: The problem solving scale is an 8-item measure assessing the degree to which youth employ skills to solve problems. All items are averaged to yield a total score that ranges from 1 = high problem solving to 4 = low problem solving; lower scores indicate a better outcome. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 556 | 591
score on a scale | 2.06 (0.40) | 2.12 (0.43)

30. Secondary Outcome: Mean Scores for Problem Solving
Description: as for outcome 29
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 559 | 587
score on a scale | 2.06 (0.42) | 2.10 (0.42)

31. Secondary Outcome: Mean Scores for Problem Solving
Description: as for outcome 29
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 564 | 584
score on a scale | 2.03 (0.40) | 2.08 (0.43)

32. Secondary Outcome: Mean Scores for Problem Solving
Description: as for outcome 29
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 562 | 581
score on a scale | 1.99 (0.39) | 2.03 (0.39)

33. Secondary Outcome: Mean Scores for Self-Esteem
Description: The self-esteem scale is a 10-item measure assessing youths' feelings of self-worth and value. All items are averaged to yield a total score that ranges from 1 = higher self-esteem to 4 = lower self-esteem; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 551 | 588
score on a scale | 2.63 (0.57) | 2.73 (0.56)

34. Secondary Outcome: Mean Scores for Self-Esteem
Description: as for outcome 33
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 553 | 582
score on a scale | 2.56 (0.57) | 2.63 (0.57)

35. Secondary Outcome: Mean Scores for Self-Esteem
Description: as for outcome 33
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 556 | 581
score on a scale | 2.49 (0.54) | 2.52 (0.58)

36. Secondary Outcome: Mean Scores for Self-Esteem
Description: as for outcome 33
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 559 | 577
score on a scale | 2.37 (0.57) | 2.42 (0.61)

37. Secondary Outcome: Mean Scores for Perceived Stress
Description: The perceived stress scale is an 8-item measure assessing the degree to which youth feel overwhelmed by stress. All items are averaged to yield a total score that ranges from 0 = low perceived stress to 5 = high perceived stress; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 566 | 604
score on a scale | 3.21 (0.66) | 3.39 (0.62)

38. Secondary Outcome: Mean Scores for Perceived Stress
Description: as for outcome 37
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 601
score on a scale | 3.19 (0.65) | 3.30 (0.64)

39. Secondary Outcome: Mean Scores for Perceived Stress
Description: as for outcome 37
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 596
score on a scale | 3.13 (0.63) | 3.19 (0.66)

40. Secondary Outcome: Mean Scores for Perceived Stress
Description: as for outcome 37
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 595
score on a scale | 3.03 (0.63) | 3.14 (0.65)

41. Secondary Outcome: Mean Scores for Coping
Description: The coping scale is a 6-item measure assessing the degree to which youth feel they can manage the difficulties in their life. All items are averaged to yield a total score that ranges from 0 = high coping skills to 3 = poor coping skills; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 563 | 603
score on a scale | 2.77 (0.45) | 2.67 (0.45)

42. Secondary Outcome: Mean Scores for Coping
Description: as for outcome 41
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 600
score on a scale | 2.75 (0.45) | 2.70 (0.47)

43. Secondary Outcome: Mean Scores for Coping
Description: as for outcome 41
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 565 | 596
score on a scale | 2.79 (0.48) | 2.74 (0.47)

44. Secondary Outcome: Mean Scores for Coping
Description: as for outcome 41
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 598
score on a scale | 2.87 (0.48) | 2.78 (0.47)

45. Secondary Outcome: Mean Scores for Peer Drug Use
Description: The peer drug use scale is a 7-item measuring that asks youth to indicate the number of close friends who have used various substances in the past month. All items are averaged to yield a total score that ranges from 0 = no peer use to 3 = all peers use; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 562 | 596
score on a scale | 0.41 (0.47) | 0.40 (0.41)

46. Secondary Outcome: Mean Scores for Peer Drug Use
Description: as for outcome 45
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 597
score on a scale | 0.51 (0.49) | 0.54 (0.48)

47. Secondary Outcome: Mean Scores for Peer Drug Use
Description: as for outcome 45
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 564 | 592
score on a scale | 0.64 (0.51) | 0.66 (0.52)

48. Secondary Outcome: Mean Scores for Peer Drug Use
Description: as for outcome 45
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 589
score on a scale | 0.74 (0.50) | 0.77 (0.53)

49. Secondary Outcome: Mean Scores for Self-Efficacy
Description: The self-efficacy scale is a 7-item measuring youths' perceived ability to handle difficult life situations. All items are averaged to yield a total score that ranges from 0 = high self-efficacy to 4 = low self-efficacy; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 556 | 585
score on a scale | 2.27 (0.51) | 2.38 (0.51)

50. Secondary Outcome: Mean Scores for Self-Efficacy
Description: as for outcome 49
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 556 | 586
score on a scale | 2.25 (0.48) | 2.36 (0.52)

51. Secondary Outcome: Mean Scores for Self-Efficacy
Description: as for outcome 49
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 561 | 589
score on a scale | 2.22 (0.47) | 2.26 (0.52)

52. Secondary Outcome: Mean Scores for Self-Efficacy
Description: as for outcome 49
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 560 | 588
score on a scale | 2.13 (0.49) | 2.19 (0.50)

53. Secondary Outcome: Mean Scores for Drug Refusal Skills
Description: The drug refusal scale is a 15-item measure assessing the likelihood of youth using various refusal strategies when offered to use alcohol, cigarettes, or marijuana. All items are averaged to yield a total score that ranges from 1 = high refusal skills to 5 = poor refusal skills; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 566 | 601
score on a scale | 1.91 (0.61) | 2.04 (0.65)

54. Secondary Outcome: Mean Scores for Drug Refusal Skills
Description: as for outcome 53
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 600
score on a scale | 1.96 (0.63) | 2.01 (0.62)

55. Secondary Outcome: Mean Scores for Drug Refusal Skills
Description: as for outcome 53
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 594
score on a scale | 1.96 (0.65) | 2.01 (0.61)

56. Secondary Outcome: Mean Scores for Drug Refusal Skills
Description: as for outcome 53
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 593
score on a scale | 1.98 (0.64) | 2.05 (0.63)

57. Secondary Outcome: Mean Scores for Assertiveness
Description: The assertiveness scale is a 3-item measure assessing how well youth believe they assert themselves. All items are averaged to yield a total score that ranges from 1 = low assertiveness to 5 = high assertiveness; higher scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 603
score on a scale | 2.83 (1.12) | 2.77 (1.11)

58. Secondary Outcome: Mean Scores for Assertiveness
Description: as for outcome 57
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 603
score on a scale | 2.92 (1.09) | 2.80 (1.11)

59. Secondary Outcome: Mean Scores for Assertiveness
Description: as for outcome 57
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 597
score on a scale | 2.92 (1.08) | 2.93 (1.11)

60. Secondary Outcome: Mean Scores for Assertiveness
Description: as for outcome 57
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 570 | 598
score on a scale | 2.97 (1.07) | 2.93 (1.10)

61. Secondary Outcome: Mean Scores for Consequences of Substance Use
Description: The consequences of substance use scale is a 13-item measure assessing how often youths' substance use has caused them trouble with the law, family, friends, and academics. All items are averaged to yield a total score that ranges from 0 = zero times to 10 = ten or more times; lower scores indicate better outcomes. The mean total score for all participants in each arm will be calculated and reported.
Time Frame: an average of 5 months from study onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 604
score on a scale | 0.08 (0.24) | 0.13 (0.41)

62. Secondary Outcome: Mean Scores for Consequences of Substance Use
Description: as for outcome 61
Time Frame: 1-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 1-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 567 | 602
score on a scale | 0.12 (0.33) | 0.13 (0.35)

63. Secondary Outcome: Mean Scores for Consequences of Substance Use
Description: as for outcome 61
Time Frame: 2-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 2-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 568 | 596
score on a scale | 0.13 (0.35) | 0.14 (0.40)

64. Secondary Outcome: Mean Scores for Consequences of Substance Use
Description: as for outcome 61
Time Frame: 3-year follow-up
Population: The analyzed population reflects only those participants who completed the assessment at 3-year follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Attention-Placebo Control
Number analyzed (Participants) | 569 | 594
score on a scale | 0.15 (0.40) | 0.13 (0.34)

ADVERSE EVENTS:
Time Frame: From enrollment to year 3 follow-up
Arm/Group | Intervention | Attention-Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/608 | 0/608
Serious Adverse Events (participants affected / at risk) | 0/608 | 0/608
Other Adverse Events (participants affected / at risk) | 0/608 | 0/608

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03954535/Prot_SAP_000.pdf